CLINICAL TRIAL: NCT06813417
Title: An Open Label Individual Patient Dose Escalation Study Investigating the Safety and Efficacy of Retreatment With GCAR1 in a Patient With Multiply Relapsed Alveolar Soft Part Sarcoma
Brief Title: CAR T Therapy With GCAR1 for Relapsed Alveolar Soft Part Sarcoma
Acronym: SPS-Q2
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health Services, Calgary (Other); Alberta Precision Laboratories (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIC-YYC-GPMB-04; HREBA.CC-24-0417 (Other: Health Research Ethics Board of Alberta)
Record Dates: First submitted 2025-01-28; First posted 2025-02-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Sarcoma; Alveolar Soft Part Sarcoma (ASPS)
Keywords: CAR T; GCAR1
MeSH Terms: conditions — Sarcoma; Sarcoma, Alveolar Soft Part

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GCAR1 (Experimental): This is an intrapatient two-dose escalation study. The patient will receive two separate intravenous infusions of cryopreserved, autologous GCAR1, with at least three months (+/- 30 days) between infusions. Both infusions will be preceded by standard lymphodepleting chemotherapy (Fludarabine 40 mg/m2 x 3 days, cyclophosphamide 600 mg/m2 x 2 days) . Dose 1 will be 5.0E6 CAR+ T cells/kg patient body weight, Dose 2 will be 2.5E7 CAR+ T cells/kg patient body weight. Infusions will be intravenous, single infusions.
  Interventions: Biological: GCAR1

INTERVENTIONS:
Biological: GCAR1 — GCAR1 is a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector encoding a chimeric antigen receptor (CAR) targeting GPNMB. The CAR comprises a single-chain variable fragment (scFv) binding domain derived from a fully human GPNMB-specific monoclonal antibody (CDX-011), a CD8 hinge and transmembrane domain, and the CD137 (4-1BB) and CD3 zeta chain intracellular signaling domains. Following infusion, the autologous GPNMB CAR T-cells expressing the genetically engineered anti-GPNMB CAR enable the specific targeting of GPNMB-expressing cells. Upon binding to GPNMB-expressing cells, the CAR transmits T cell activation signals that promote the elimination of target cells through CAR T cell degranulation and the release of cytotoxic molecules. The cellular signal also facilitates CAR T cell proliferation and persistence that may enable prolonged disease control through immunosurveillance3.

SUMMARY:
A single patient study to determine whether GCAR1 is safe and effective for re-treatment of alveolar soft part sarcoma (ASPS) with GPNMB surface expression that has relapsed and is not responding to usual treatment.

DETAILED DESCRIPTION:
CLIC-YYC-GPNMB-04 is an Open Label Individual Patient (OLIP)/Single Patient Study (SPS) developed according to the Health Canada template and guidelines released in 2019 for studies to access therapies not otherwise available to patients, in the situation where there are no options of treatment or cure remaining. The patient under consideration for CLIC-YYC-GPNMB-04 has refractory, progressive metastatic alveolar soft part sarcoma (ASPS). There are no standard therapies for relapsed ASPS known to provide potential for cure, and there are no clinical trials available in Canada for consideration. We propose to re-treat the patient with GCAR1, a patient-specific cell therapy product containing a mixture of autologous lymphocytes transduced with a lentiviral vector containing a chimeric antigen receptor (CAR) that enables the specific targeting towards tumor cells expressing the cell surface protein glycoprotein non-metastatic B (GPNMB). The patient was previously treated with GCAR1 under CLIC-YYC-GPNMB-01 (c#276646).

ELIGIBILITY:
Inclusion Criteria:

* The patient must provide informed consent
* Adequate organ function, defined as creatinine clearance >30 ml/min and LVEF >45%

Exclusion Criteria:

* Any active uncontrolled infection
* Pregnancy or nursing
* Anti-cancer therapy within 21 calendar days prior to the first dose of lymphodepleting chemotherapy. If subject has received anti-cancer therapy, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy as per the discretion of the Qualified Investigator/Co-Investigator

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2030-01-30 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | Diagnostic imaging (CT and/or MRI) will be performed at baseline (pre-treatment) and then subsequently at 4-6 weeks after GCAR1 infusion, and at 3 months, 6 months, 9 months and 1 year after last infusion to evaluate response to therapy.
  The overall response assessment considers the response of the target and non-target lesions and development of new lesions.
  Response Classification of Target Lesions, CNS lesions and Non-Target Lesions
  * Complete response (CR):
  * Partial response (PR):
  * Progressive disease (PD):
  * Stable disease (SD):

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada